CLINICAL TRIAL: NCT05232487
Title: Comparison of Swiss Versus Standard Low Back Acupuncture in Patients With Chronic Low Back Pain. A Randomized, Controlled, Single-blind, Monocentric Clinical Study
Brief Title: Comparison of Swiss Versus Standard Low Back Acupuncture in Patients With Chronic Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Li Yiming (Other)
Collaborators: Swiss University for Traditional Chinese Medicine (Unknown)
Responsible Party: Sponsor-Investigator, Li Yiming, Yiming Li, Prof. Dr. TCM univ. (CN) Dr. med., TCM Ming Dao
Organization: TCM Ming Dao (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Study ID: TCM_AKU01/2021
Record Dates: First submitted 2021-12-30; First posted 2022-02-09 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Chronic Low-back Pain
Keywords: chronic low back pain; Acupuncture; Standard acupuncture; Swiss low back acupuncture

STUDY DESIGN:
Intervention Model Description: This study is a randomized, controlled, single-blind, parallel trial, allocating patients with CLBP 1:1 to either 9 weeks of SLBA or SA therapy.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients will be randomized by using the web-based secuTrial randomization tool and by applying an allocation ratio of 1:1 to SLBA and SA therapy. Patients and data analysts will be blinded to the intervention (SLBA or SA), however, acupuncturists performing the acupuncture sessions will not be blinded to the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Swiss low back acupuncture group (Experimental): Participants in this group will be treated with the Swiss low back acupuncture method.
  Interventions: Other: Swiss low back acupuncture (SLBA)
- Standard acupuncture group (Active Comparator): Participants in this group will be treated with the standard acupuncture method.
  Interventions: Other: Standard acupuncture (SA)

INTERVENTIONS:
Other: Swiss low back acupuncture (SLBA) — Participants are placed in the prone position (if required with a pillow under the abdomen). Then acupuncture is applied to the back of the body. The treatment takes place for the duration of 9 weeks (2x per week from week 1 to 6 and 1x a week from week 7 to 9). One treatment session lasts about 50-60 minutes.
  Swiss low back pain acupuncture The SLBA method is a further developed method from the Jiu Gong acupuncture technique, also known as the Nine Palace-Points on the spine. The following acupuncture points will be used: LV3/ LV5, Tai Xi (Kl 3), Fe Yang (BL 58), Tai Chong (LR 3), Guang Ming (GB 37), Tai Xi (Kl 3) and Fe Yang (BL 58).
  Arms: Swiss low back acupuncture group
Other: Standard acupuncture (SA) — Participants are placed in the prone position (if required with a pillow under the abdomen). Then acupuncture is applied to the back of the body. The treatment takes place for the duration of 9 weeks (2x per week from week 1 to 6 and 1x a week from week 7 to 9). One treatment session lasts about 50-60 minutes. The SA method is described in the acupuncture textbook for TCM in China and all acupuncture points are selected based on TCM principles, international literature, and the opinion of national and international TCM experts. The following points have been selected: Ming Men (GV 4), Zhi Shi (BL 52), Tai Xi (KI 3) Yao Guan (GV 3), Guan Yuan Shu (BL 26), Ge Shu (BL 17), Ci Liao (BL 32), Wei Zhong (BL 40), Ji Zhong (GV 6), Yao Yang Guan (GV 3), Shen Shu (BL 23), Da Chang Shu (BL 25) and A-Shi points.
  Arms: Standard acupuncture group

SUMMARY:
Low back pain (LBP) is very common, widespread, and represents a multidimensional syndrome. It affects physical activity and function, health-related quality of life, and employment status. The lifetime prevalence of acute low back pain is approximately 80%. The prevalence of chronic low back pain (CLBP) in the general population is reported to be 8% to 21%. Several clinical trials have provided evidence to support the efficacy of acupuncture in the treatment of LBP, however, the optimal acupuncture treatment for CLBP has not been extensively studied.

DETAILED DESCRIPTION:
Low back pain (LBP) is a common, widespread and multifaceted syndrome and represents one of the leading sources of years lived with disability. In Switzerland, patients with LBP generated mean annual costs of 467 million Euro in 2016 and 2017, respectively. Moreover, quantity of prescriptions per patient was reported to be 5 - 6 per year, causing pain medication costs of 4.7 million Euro. It is estimated that 20% of acute LBP can manifest as chronic LBP (CLBP), defined as pain lasting longer than three months. CLBP does not only negatively impact the quality of life, functional status, and working capability of those suffering, but also plays a pivotal role of the large annual health care costs for LBP in Switzerland and worldwide. Pharmacological therapies with at least a small magnitude of effect for pain relief in CLBP include non-steroidal anti-inflammatory drugs, opioids, Tramadol and antidepressants. Additionally, non-pharmacological therapies with at least a small magnitude of effect for pain relief in CLBP include exercise, motor control exercise, Yoga, mindfulness-based stress reduction, electromyography biofeedback, cognitive-behavioral therapy, multidisciplinary rehabilitation and acupuncture.

In this context and during the last decades and centuries, different acupuncture methods evolved, among others, the acupuncture method newly termed "Swiss low back acupuncture" (SLBA). The SLBA originates from Jiu Gong Points (九宫穴), which is the abbreviation for "Nine Spinal Points" (脊椎九宫穴). The particular sites of Jiu Gong Points were evolved from the eight trigrams and nine palaces square (Ba Gua Jiu Gong fang 八卦九宫方). The eight trigrams (Ba Gua 八卦) are a set of metaphysical and philosophical sigmas composed of three components of yin and yang, which are the essential concept of all-natural phenomena. Nine palaces (Jiu Gong, 九宫), an element of the eight trigrams, correspond to the nine regions in ancient China (Jiu Ye, 九野). They represent the four main (North=kidney; South=heart; East=liver; West=lung; Earth=spleen) and four secondary cardinal points and the earth as the center. In 825 patients with LBP due to lumbar herniated disc, it has been shown that hot needle acupuncture (热针) using Jiu Gong Points around the most significant lesion of the lumbar vertebrae results in good improvements of pain. The uncontrolled study reported a cure of LBP in 65.2% of cases and an improvement of clinical symptoms of 32.4%. Due to the positive report, the hot needle acupuncture using Jiu Gong Points has further evolved in Switzerland and might be a promising tool to treat CLBP, since the optimal method of acupuncture against CLBP remains to be elucidated. However, the efficacy of SLBA has never been quantitatively compared to SA and a randomized clinical trial is warranted to provide first robust evidence on its performance in CLBP.

Therefore, the purpose of this study is to conduct the first randomized clinical trial comparing SLBA and SA on pain relief in patients with CLBP.

ELIGIBILITY:
Inclusion Criteria:

* Female and male participants;
* Age between 18 and 75 years;
* Clinical diagnosis of CLBP with a disease duration of more than 3 months and an average pain intensity of minimally 4 points on a 11-point pain-numerical rating scale (pain-NRS) on the previous 7 days;
* Sufficient knowledge of German to complete the questionnaires.

Exclusion Criteria:

* All participants who do not meet the above-mentioned inclusion criteria;
* History or known severe concomitant diseases (e.g. abdominal aortic aneurysm, heart disease, cancer, psychiatric disorders).
* Other causes of low back pain not related to the clinical diagnosis of CLBP including inflammatory, malignant, or autoimmune disease;
* Planned or previous back surgery within 6 months
* Use of corticosteroids and/or other pain-relieving drugs that act through the central nervous system;
* Initiation of another therapy for CLBP within the last 4 weeks, e.g. physiotherapy;
* Preceding acupuncture treatment for CLBP during the past 6 months;
* Pregnancy;
* Participation in another clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Pain Severeity rated by 11-Point Numerical Rating Scale | Difference in change between 9 weeks of treatment with SLBA compared to SA therapy.
  Pain severity will be assessed by the 11-point numerical rating scale, ranging from 0 "No pain" to 10 "maximal pain".

SECONDARY OUTCOMES:
Changes in biopsychosocial health and quality of life | Difference in change between 9 weeks of treatment with SLBA compared to SA therapy; after 3 and 6 months follow-up.
  The Short Form 36 will be assessed at the start of the intervention (T1) and after completion of the last intervention (T2), as well as at follow-up (3 months after the end of intervention [T3] / 6 months after the end of intervention [T4]).
Changes in symptomatic distress | Difference in change between 9 weeks of treatment with SLBA compared to SA therapy; after 3 and 6 months follow-up.
  The SCL-90 R. Scales of Anxiety (10 items), Depression (13 items), and Somatization (12 items) will be assessed at the start of the intervention (T1) and after completion of the last intervention (T2), as well as at follow-up (3 months after the end of intervention [T3] / 6 months after the end of intervention [T4]).
Changes in functional status and disability | Difference in change between 9 weeks of treatment with SLBA compared to SA therapy; after 3 and 6 months follow-up.
  The score of the Oswestry Disability Index will be assessed at the start of the intervention (T1) and after completion of the last intervention (T2), as well as at follow-up (3 months after the end of intervention [T3] / 6 months after the end of intervention [T4]).
Multidimensional Pain Inventory (MPI) - pain severity score | Difference in change between 9 weeks of treatment with SLBA compared to SA therapy.
  Pain severity score will be calculated from 3 items:
  * Rate the severity of your current pain (now, at the moment).
  * How severe was your pain in the last week? (average)
  * How much do you suffer from your pain?
  The total score will be transformed into 0 (maximal pain) to 100 points (no pain) by the following equation: 100 - (scored points)/18 ×100
  MPI will be assessed at the start of the intervention (T1) and after completion of the last intervention (T2), as well as at follow-up (3 months after the end of intervention [T3] / 6 months after the end of intervention [T4]).
Pain diary | During the 9 weeks of treatment with SLBA compared to SA therapy.
  Patients will be asked to complete a daily pain diary during the 9-weeks of acupuncture therapy (completed at the end of each day, before going to bed). In this diary, the patients will rate their perceived pain severity from 0 (none) to 5 (almost intolerable pain) during pre-defined periods of the day. Furthermore, drug intake related to pain relief will be documented.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Furain, PhD, Principal Investigator — Swiss University for Traditional Chinese Medicine
Locations (1):
- Swiss TCM UNI, Bad Zurzach, Canton of Aargau, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with an academic interest in LBP. Data or samples shared will be coded, with no Protected Health Information included. Approval of the request and execution of all applicable agreements are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data requests can be submitted starting 12 months after article publication, and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact: michael.furian@usz.ch

REFERENCES:
- [Background] Angst F, Verra ML, Lehmann S, Aeschlimann A. Responsiveness of five condition-specific and generic outcome assessment instruments for chronic pain. BMC Med Res Methodol. 2008 Apr 25;8:26. doi: 10.1186/1471-2288-8-26. PMID 18439285
- [Background] Angst F, Verra ML, Lehmann S, Aeschlimann A, Angst J. Refined insights into the pain-depression association in chronic pain patients. Clin J Pain. 2008 Nov-Dec;24(9):808-16. doi: 10.1097/AJP.0b013e31817bcc5f. PMID 18936599
- [Background] Benz T, Lehmann S, Elfering A, Sandor PS, Angst F. Comprehensiveness and validity of a multidimensional assessment in patients with chronic low back pain: a prospective cohort study. BMC Musculoskelet Disord. 2021 Mar 20;22(1):291. doi: 10.1186/s12891-021-04130-x. PMID 33743669
- [Background] Chan MWC, Wu XY, Wu JCY, Wong SYS, Chung VCH. Safety of Acupuncture: Overview of Systematic Reviews. Sci Rep. 2017 Jun 13;7(1):3369. doi: 10.1038/s41598-017-03272-0. PMID 28611366
- [Background] Hasenbring, M. (2004). Rückenschmerzen: Der Chronifizierung frühzeitig entgegenwirken. In Neuroorthopädie (pp. 13-21). Steinkopff. https://doi.org/10.1007/978-3-7985-1949-7_3
- [Background] Kim J, Shin W. How to do random allocation (randomization). Clin Orthop Surg. 2014 Mar;6(1):103-9. doi: 10.4055/cios.2014.6.1.103. Epub 2014 Feb 14. PMID 24605197
- [Background] Labots G, Jones A, de Visser SJ, Rissmann R, Burggraaf J. Gender differences in clinical registration trials: is there a real problem? Br J Clin Pharmacol. 2018 Apr;84(4):700-707. doi: 10.1111/bcp.13497. Epub 2018 Feb 12. PMID 29293280
- [Background] Lee CP, Fu TS, Liu CY, Hung CI. Psychometric evaluation of the Oswestry Disability Index in patients with chronic low back pain: factor and Mokken analyses. Health Qual Life Outcomes. 2017 Oct 3;15(1):192. doi: 10.1186/s12955-017-0768-8. PMID 28974227
- [Background] Leem J. Does acupuncture increase the risk of bleeding in patients taking warfarin? Integr Med Res. 2015 Jun;4(2):119-121. doi: 10.1016/j.imr.2015.04.001. Epub 2015 Apr 22. No abstract available. PMID 28664117
- [Background] Mcculloch M, Nachat A, Schwartz J, Casella-Gordon V, Cook J. Acupuncture safety in patients receiving anticoagulants: a systematic review. Perm J. 2015 Winter;19(1):68-73. doi: 10.7812/TPP/14-057. Epub 2014 Nov 24. PMID 25432001
- [Background] Mu J, Furlan AD, Lam WY, Hsu MY, Ning Z, Lao L. Acupuncture for chronic nonspecific low back pain. Cochrane Database Syst Rev. 2020 Dec 11;12(12):CD013814. doi: 10.1002/14651858.CD013814. PMID 33306198
- [Background] Pignon JP, Arriagada R. Early stopping rules and long-term follow-up in phase III trials. Lung Cancer. 1994 Mar;10 Suppl 1:S151-9. doi: 10.1016/0169-5002(94)91677-2. PMID 8087505
- [Background] Salaffi F, Stancati A, Silvestri CA, Ciapetti A, Grassi W. Minimal clinically important changes in chronic musculoskeletal pain intensity measured on a numerical rating scale. Eur J Pain. 2004 Aug;8(4):283-91. doi: 10.1016/j.ejpain.2003.09.004. PMID 15207508
- [Background] Schmitz N, Hartkamp N, Kiuse J, Franke GH, Reister G, Tress W. The Symptom Check-List-90-R (SCL-90-R): a German validation study. Qual Life Res. 2000 Mar;9(2):185-93. doi: 10.1023/a:1008931926181. PMID 10983482
- [Background] Witt CM, Pach D, Brinkhaus B, Wruck K, Tag B, Mank S, Willich SN. Safety of acupuncture: results of a prospective observational study with 229,230 patients and introduction of a medical information and consent form. Forsch Komplementmed. 2009 Apr;16(2):91-7. doi: 10.1159/000209315. Epub 2009 Apr 9. PMID 19420954
- [Background] Vickers AJ, Vertosick EA, Lewith G, MacPherson H, Foster NE, Sherman KJ, Irnich D, Witt CM, Linde K; Acupuncture Trialists' Collaboration. Acupuncture for Chronic Pain: Update of an Individual Patient Data Meta-Analysis. J Pain. 2018 May;19(5):455-474. doi: 10.1016/j.jpain.2017.11.005. Epub 2017 Dec 2. PMID 29198932
- [Background] von der Heyde, R. (2007). Assessment of Functional Outcomes. In Fundamentals of Hand Therapy (pp. 98-113). Elsevier. https://doi.org/10.1016/B0-32-303386-5/50009-6
- [Background] Xiang Y, He JY, Tian HH, Cao BY, Li R. Evidence of efficacy of acupuncture in the management of low back pain: a systematic review and meta-analysis of randomised placebo- or sham-controlled trials. Acupunct Med. 2020 Feb;38(1):15-24. doi: 10.1136/acupmed-2017-011445. Epub 2019 Sep 16. PMID 31526013
- [Derived] Pradhan SK, Angst F, Xu J, Gantenbein AR, Lehmann S, Sandor PS, Li Y, Furian M. Comparison of Swiss versus Standard Acupuncture in Patients with Chronic Low Back Pain. A Study Protocol for a Randomized, Controlled, Single-Blind, Parallel Trial. J Pain Res. 2022 Dec 22;15:4055-4064. doi: 10.2147/JPR.S388558. eCollection 2022. PMID 36579179